CLINICAL TRIAL: NCT04422158
Title: Impact of Nuun Electrolyte Tablets on Hydration Status in Active Men and Women: Single-blinded Study
Brief Title: Impact of Nuun Electrolyte Tablets on Hydration Status in Active Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Nuun & Company, Inc (Nuun) (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of School of Health Studies, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2020-327
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hydration
Keywords: electrolyte
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, placebo-controlled, cross-over with non-directional hypothesis regarding the potential differences between the two different dosages tested.
Who Masked: Participant
Masking Description: Drinks will be prepared without subjects aware of which drink they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nuun Single strength (Experimental): 3 Nuun electrolyte tablets will be dissolved in 1.4 liters of water. Subjects will drink one liter of the prepared solution over 30 min (250 mL every 7.5 min)
  Interventions: Dietary Supplement: Nuun electrolyte tablet; Other: water
- Nuun Double strength (Experimental): 6 Nuun electrolyte tablets will be dissolved in 1.4 liters of water. Subjects will drink one liter of the prepared solution over 30 min (250 mL every 7.5 min)
  Interventions: Dietary Supplement: Nuun electrolyte tablet; Other: water
- Control (Placebo Comparator): Subjects will drink one liter of water over 30 min (250 mL every 7.5 min)
  Interventions: Other: water

INTERVENTIONS:
Dietary Supplement: Nuun electrolyte tablet — Each table contains 2 grams of carbohydrate and a combination of electrolytes. calcium (13mg, 1%DV), sodium (300mg, 13%DV), potassium (150mg, 3%DV), magnesium (25mg, 6%DV), and chloride (40mg, 2%DV).
  Arms: Nuun Double strength; Nuun Single strength
Other: water — water

SUMMARY:
The purpose of this study is to determine the impact of Nuun electrolyte tablets on hydration status in young and active men and women. We will follow a similar approach as used by Maughan and colleagues (2016) to measure the beverage hydration index (the relative amount of urine passed after consumption of a drink compared to water). It is hypothesized that Nuun electrolyte tablets will result in a greater hydration status as compared to water only. Due to the fact that athletes use Nuun tablets at varying dosages, we will evaluate Nuun at both a single dosage and a double dosage. We maintain a non-directional hypothesis regarding the potential differences between the two different dosages tested.

DETAILED DESCRIPTION:
Maintaining adequate hydration is essential to optimal health and athletic performance. When individuals exercise (in particular in a warm environment), they can lose excessive amounts of fluids through sweating, along with necessary electrolytes (e.g., sodium, potassium, chloride). With dehydration, individuals may feel sluggish and can experience impaired physical performance.

Many attempts have been made to improve and measure the hydration status of active individuals. This typically involves the ingestion of fluids leading up to activity (typically plain water), as well as the ingestion of fluids during the activity itself (water, along with a diluted carbohydrate/electrolyte beverage). This approach seems to work well; however, some debate remains over what the best fluid is to consume, in particular related to the macronutrient type and the specific electrolyte mix.

Related to the above, it is well-accepted that electrolyte replenishment is of importance, both during and following exercise-to aid in rehydration for subsequent bouts. The use of electrolytes (sodium in particular) has been used for decades to aid athlete hydration and has led to the development of various sport drinks-which also include small amounts of carbohydrate. However, one problem with carbohydrate ingestion is that some individuals experience gastrointestinal (GI) upset following carbohydrate ingestion before and during an event, despite very good physical performance outcomes. Due to this GI upset, some individuals (in particular recreationally active individuals who are not competing at high levels) rely solely on water and seek a method to ingest the lost electrolytes. In addition, some individuals prefer to have both plain water and an electrolyte beverage during their training/competition sessions and in some activities (e.g., running, cycling), carrying multiple bottles of fluid is difficult.

The solution to the above issues for many athletes is the use of electrolyte tablets. These can be dropped into plain water and will dissolve into a flavored electrolyte-rich beverage. They are easy to transport and provide the needed electrolytes to replace those that are lost through intense and/or long duration exercise.

Nuun electrolyte tablets provide only 2 grams of carbohydrate and a combination of electrolytes, provided at a relatively low percentage of the Daily Value (DV). The DV tells us how much a particular nutrient in a serving of a food product contributes to a daily diet, based on a standard 2000 calorie diet. Nuun tablets contain: calcium (13mg, 1%DV), sodium (300mg, 13%DV), potassium (150mg, 3%DV), magnesium (25mg, 6%DV), and chloride (40mg, 2%DV). These tablets contain a small percentage of the needed total electrolytes but adequate amounts to replace lost electrolytes as a result of physical activity.

While Nuun tablets are commercially available and have received positive reviews from end users, there have been no studies to date to evaluate the impact of these tablets on hydration status. Therefore, the purpose of this study is to determine the impact of Nuun electrolyte tablets on hydration status in young and active men and women. We will follow a similar approach as used by Maughan and colleagues to measure the beverage hydration index (the relative amount of urine passed after consumption of a drink compared to water). It is hypothesized that Nuun electrolyte tablets will result in a greater hydration status as compared to water only. Due to the fact that athletes use Nuun tablets at varying dosages, we will evaluate Nuun at both a single dosage and a double dosage. We maintain a non-directional hypothesis regarding the potential differences between the two different dosages tested.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 29.9 kg/m2 (not obese)
* Consumes 2 liters of water daily
* Exercised 3 hours/week over the past 6 months

Exclusion Criteria:

* Obese
* Pregnant or trying to become pregnant
* Tobacco user
* Cardiac Disease
* Consumed alcohol within 48 hours of testing visit
* Consumed caffeine within 48 hours of testing visit
* Strenuous excercise 24 hours prior to testing visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Body weight | baseline
  Body weight will be measured
Body weight | 4 hours after drink consumption
  Body weight will be measured
Urine volume | Immediately after completing intervention
  Volume of urine output will be measured
Urine volume | 1 hour after intervention
  Volume of urine output will be measured
Urine volume | 2 hours after intervention
  Volume of urine output will be measured
Urine volume | 3 hours after intervention
  Volume of urine output will be measured
Urine volume | 4 hours after intervention
  Volume of urine output will be measured
Urine mass | Immediately after completing intervention
  Urine output will be measured using a scale
Urine mass | 1 hour after intervention
  Urine output will be measured using a scale
Urine mass | 2 hours after intervention
  Urine output will be measured using a scale
Urine mass | 3 hours after intervention
  Urine output will be measured using a scale
Urine mass | 4 hours after intervention
  Urine output will be measured using a scale
Blood Pressure | at baseline
  Blood pressure will be measured.
Blood Pressure | 1 hour after intervention
  Blood pressure will be measured.
Blood Pressure | 2 hours after intervention
  Blood pressure will be measured.
Blood Pressure | 3 hours after intervention
  Blood pressure will be measured.
Blood Pressure | 4 hours after intervention
  Blood pressure will be measured.
Heart Rate | baseline
  Heart Rate will be measured
Heart Rate | 1 hour after intervention
  Heart Rate will be measured
Heart Rate | 2 hours after intervention
  Heart Rate will be measured
Heart Rate | 3 hours after intervention
  Heart Rate will be measured
Heart Rate | 4 hours after intervention
  Heart Rate will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No